CLINICAL TRIAL: NCT03596567
Title: A PHASE 1, OPEN-LABEL, SINGLE DOSE, PARALLEL GROUP STUDY TO EVALUATE THE PHARMACOKINETICS OF GLASDEGIB (PF-04449913) IN SUBJECTS WITH IMPAIRED RENAL FUNCTION
Brief Title: Glasdegib Renal Impairment Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B1371017
Record Dates: First submitted 2018-04-02; First posted 2018-07-24 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Renal Impairment
Keywords: Glasdegib; PF-04449913; Pharmacokinetics; Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Normal Renal Function Group (Experimental): Subjects with estimated glomerular filtration rate (eGFR) of => 90 ml/min
  Interventions: Drug: Glasdegib single 100 mg dose in normal healthy subjects
- Moderate Renal Impairment Group (Experimental): Subjects with estimated glomerular filtration rate (eGFR) of => 30ml/min and < 60 ml/min
  Interventions: Drug: Glasdegib single 100 mg dose in moderate renal impairment subjects
- Severe Renal Impairment Group (Experimental): Subjects with estimated glomerular filtration rate (eGFR) of < 30 ml/min and not requiring dialysis
  Interventions: Drug: Glasdegib single 100 mg dose in severe renal impairment subjects

INTERVENTIONS:
Drug: Glasdegib single 100 mg dose in normal healthy subjects — A single dose of 100 mg glasdegib tablet will be administered after an overnight fast, followed by serial PK collection, discharge and follow -up.
  Arms: Normal Renal Function Group
Drug: Glasdegib single 100 mg dose in moderate renal impairment subjects — A single dose of 100 mg glasdegib tablet will be administered to subjects with moderate renal impairment, after an overnight fast, followed by serial PK collection, discharge and follow -up.
  Arms: Moderate Renal Impairment Group
Drug: Glasdegib single 100 mg dose in severe renal impairment subjects — A single dose of 100 mg glasdegib tablet will be administered to subjects with severe renal impairment, after an overnight fast, followed by serial PK collection, discharge and follow -up.
  Arms: Severe Renal Impairment Group

SUMMARY:
The goal of this study is to administer single dose (100 mg) glasdegib tablet to subjects with normal, moderate and severe renal impairment and estimate the effect, if any, of this renal impairment on glasdegib pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects of non child bearing potential and/or male subjects who, at the time of screening, are between the ages of 18 and 75 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG or clinical laboratory tests.
2. Female subjects of nonchildbearing potential must meet at least 1 of the following criteria:

   1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; with a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state;
   2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
   3. Have medically confirmed ovarian failure. All other female subjects (including females with tubal ligations) are considered to be of childbearing potential.
3. Body mass index (BMI) of 17.5 to 40 kg/m2; and a total body weight >50 kg (110 lb).
4. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
5. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Subjects with Normal Renal Function will Need to Meet the Following Criteria in addition -

1. Normal renal function, eGFR=>90 mL/min, based on the MDRD equation.
2. Matched for age (+/-10years) weight +/-15kg, and gender to subjects in the impaired renal function groups

Subjects with Impaired Renal Function will Need to Meet the Following Criteria in Addition to Those Above

1. Good general health commensurate with the population with chronic kidney disease (renal impairment). 'Health' is defined as no clinically relevant abnormalities (with the exception of hypertension, diabetes mellitus, hyperparathyroidism, ischemic heart disease, etc. as long as, in the opinion of the investigator, the subject is medically stable, is on a stable drug regimen and can abide by the meals and dietary restrictions outlined in protocol identified by a detailed medical history, full physical examination, measurement of pulse rate and 12 lead ECG as well as clinical laboratory tests (except serum creatinine and eGFR).
2. Stable drug regimen defined as not starting a new drug or changing dosage within seven days or five half lives (whichever is longer) before dosing the study drug.
3. Any form of renal impairment except acute nephritic syndrome (subjects with history of previous nephritic syndrome but in remission can be included).
4. Meet one of the following eGFR criteria during the screening period based on the MDRD equation:

   1. Moderate renal impairment: eGFR 30 mL/min and <60 mL/min, or
   2. Severe renal impairment: eGFR <30 mL/min, but not requiring hemodialysis. For subjects in all groups, the values of serum creatinine obtained at the two screening visits should not be more than 20% different.

      Exclusion Criteria:

      -Any condition possibly affecting drug absorption (eg, gastrectomy, achlorhydria).

      Renal allograft recipients

      Urinary incontinence without catheterization.

      Concurrent use of any of the following food or drugs known to inhibit CYP3A4 (consult the Sponsor if in doubt whether a food or a drug falls into any of the above categories) within 7 days or 5 half lives (whichever is longer) prior to the dose of glasdegib, until the completion of the last PK sample collection.

      Concurrent use of any of the following food or drugs known to induce CYP3A4 (consult the Sponsor if in doubt whether a food or a drug falls into any of the above categories) within 12 days or 5 half lives (whichever is longer) prior to the first dose of trial medication until the completion of the last PK sample collection.

      Pregnant female subjects; breastfeeding female subjects; fertile male subjects who are unwilling or unable to use two highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 90 days after the last dose of investigational product and, refrain from sperm donation for the duration of the Study and for at least 90 days after the last dose of investigational product.

      Subjects with ANY of the following abnormalities in clinical laboratory tests at Screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:
      * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level > upper limit of normal (ULN);
      * Total bilirubin level 1.5 × ULN; subjects with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is not greater than 0.5 mg/dL.

      For subjects with renal impairment, the following important additional criteria are:

      Subjects with other clinically significant disease that may affect the safety of the subject or that may affect the pharmacokinetics of glasdegib (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing). Subjects with any significant hepatic, cardiac, or pulmonary disease or subjects who are clinically nephrotic. Hypertension, diabetes mellitus, hyperparathyroidism, ischemic heart disease, etc is not cause for exclusion as long as the subject is medically stable and any drugs that are administered for these conditions are not expected to interfere with the pharmacokinetics of glasdegib.

      Screening blood pressure =>180mm Hg (systolic) or>=110 mm Hg (diastolic), following at least 5 minutes of supine rest. If initial blood pressure (BP) is 180 mm Hg (systolic) or 110 mm Hg (diastolic), the BP should be repeated two more times and the average of the three BP values should be used to determine the subject's eligibility.

      Screening supine 12 lead ECG demonstrating QTcF >470 msec or a QRS interval >120 msec. If initial QTcF exceeds 470 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTcF or QRS values should be used to determine the subject's eligibility.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 6 days
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 6 days
  AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]). | 34 days
  concomitant medication and adverse event monitoring.
PR/ECGs | 34 days
  PR interval (msec),
Hematology Lab Panel | 34 days
  Platelet count (10^3/mm^3)
BUN /Chemistry Lab Panel | 34 days
  BUN (mg/dL)
pH/Urinalysis Lab Panel | 34 days
  pH (no unit)
Blood Pressure | 34 days
  Supine Systolic and Diastolic blood pressure (mm of Hg). Reported as Systolic/Diastolic
Pulse Rate | 34 days
  Pulse Rate will be reported in beats per minute.
ECGs | 34 days
  Heart Rate (beats per minute)
Hemoglobin /Hematology Lab Panel | 34 days
  Hemoglobin (g/dL)
Hematology Lab Panel | 34 days
  Hematocrit (%)
Hematology Lab Panel | 34 days
  RBC Count (10^6/mm^3)
Hematology Lab Panel | 34 days
  MCV (femto Liters)
Hematology Lab Panel | 34 days
  MCH (pictograms/cell)
Potassium/Chemistry Lab Panel | 34 days
  Potassium (Meq/L)
AST/Chemistry Lab Panel | 34 days
  AST (U/L)
Albumin/Chemistry Lab Panel | 34 days
  Albumin (g/dL)
MCHC/Hematology Lab Panel | 34 days
  MCHC (10^3/mm^3)
WBC count/Hematology Lab Panel | 34 days
  WBC count (10^3/mm^3),
Total neutrophils/Hematology Lab Panel | 34 days
  Total neutrophils (Abs)(10^3/mm^3),
Eosinophils/Hematology Lab Panel | 34 days
  Eosinophils (Abs)(10^3/mm^3
Monocytes/Hematology Lab Panel | 34 days
  Monocytes (Abs)(10^3/mm^3)
Basophils/Hematology Lab Panel | 34 days
  Basophils (Abs) (10^3/mm^3)
Lymphocytes/Hematology Lab Panel | 34 days
  Lymphocytes (Abs) (10^3/mm^3)
Total Protein/Chemistry Lab Panel | 34 days
  Total Protein (g/dL)
ALT/Chemistry Lab Panel | 34 days
  ALT (U/L)
Alkaline Phosphate/Chemistry Lab Panel | 34 days
  Alkaline Phosphate (U/L)
Sodium/Chemistry Lab Panel | 34 days
  Sodium (Meq/L)
Chloride/Chemistry Lab Panel | 34 days
  Chloride (Meq/L)
Creatinine/Chemistry Lab Panel | 34 days
  Creatinine (mg/dL),
Glucose/Chemistry Lab Panel | 34 days
  Glucose (mg/dL),
Calcium/Chemistry Lab Panel | 34 days
  Calcium (mg/dL),
Total Bilirubin/Chemistry Lab Panel | 34 days
  Total Bilirubin (mg/dL),
Uric acid/Chemistry Lab Panel | 34 days
  Uric acid (mg/dL)
Magnesium/Chemistry Lab Panel | 34 days
  Magnesium (mg/dL)
QTc/ECGs | 34 days
  QTc interval (msec)
QRS/ECGs | 34 days
  QRS interval (msec)
Glucose/Urinalysis Lab Panel | 34 days
  Glucose (qual) (no unit)
Protein/Urinalysis Lab Panel | 34 days
  Protein (qual) (no unit)
Blood/Urinalysis Lab Panel | 34 days
  Blood (qual) (no units)
Ketones/Urinalysis Lab Panel | 34 days
  Ketones (no units)
Nitrites/Urinalysis Lab Panel | 34 days
  Nitrites (no units)
Leukocyte /Urinalysis Lab Panel | 34 days
  Leukocyte esterase (no units)
Urobilinogen/Urinalysis Lab Panel | 34 days
  Urobilinogen (no unit)
Urine bilirubin/Urinalysis Lab Panel | 34 days
  Urine bilirubin (no unit)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - University of Miami Division of Clinical Pharmacology, Miami, Florida
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Prism Clinical Research LLC, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Shaik N, LaBadie RR, Hee B, Chan G. Evaluation of the impact of renal impairment on the pharmacokinetics of glasdegib in otherwise healthy volunteers. Cancer Chemother Pharmacol. 2021 Feb;87(2):241-250. doi: 10.1007/s00280-020-04207-9. Epub 2021 Jan 3. PMID 33388951
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1371017